CLINICAL TRIAL: NCT07162129
Title: Online Transdiagnostic Group Cognitive Behavioural Therapy (CBT) for Postpartum Depression and Anxiety: A Pilot Randomized Controlled Trial
Brief Title: Online Transdiagnostic Group CBT for Postpartum Depression and Anxiety
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Group CBT for PPD & PPA Pilot
Record Dates: First submitted 2025-08-29; First posted 2025-09-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression (PPD); Postpartum Anxiety
Keywords: Transdiagnostic; Postpartum Depression; Postpartum Anxiety; Cognitive Behavioural Therapy
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy; Tuberculin

STUDY DESIGN:
Intervention Model Description: A parallel-group Ontario-wide RCT with experimental (CBT group) and TAU (control) groups will address our objectives. Participants will be randomly assigned in a 1:1 ratio to the treatment or control groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and the research coordinator cannot be blinded to group condition though the research assistants making reminder calls and data analysts will not be aware of group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-week Transdiagnostic Group CBT Intervention (Experimental): The experimental group will receive a 10-week transdiagnostic group CBT intervention delivered by a pair of trained mental health providers (psychiatrists, psychologists, social workers, nurses and/or registered psychotherapists) in addition to receiving treatment as usual.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Postpartum Depression (PPD) and Anxiety
- Control - usual care (No Intervention): Participants randomized to the No Intervention group will continue to receive treatment as usual (standard postnatal care). A list of resources will be emailed.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Postpartum Depression (PPD) and Anxiety — Cognitive Behavioral Therapy (CBT) is a type of psychotherapy (talk therapy). Each session will be two hours in duration. The 1st hour involves teaching and practice of CBT skills followed by one hour of unstructured discussion about topics relevant to PPD and PPA (sleep, supports, transitions). Each group will be delivered online via Zoom and guided by our intervention manual.
  Arms: 10-week Transdiagnostic Group CBT Intervention

SUMMARY:
The purpose of this pilot study is to test the feasibility of an online 10-Week group cognitive behavioural therapy (CBT; a type of talking therapy) intervention for postpartum depression and anxiety that is led by psychotherapists, social workers, a psychologist and/or a psychiatrist. Mothers and birthing parents who are 18 years or older, have an infant under 12 months, living in Ontario and who have postpartum depression and/or anxiety symptoms will be assigned with a 50/50 chance (like flipping a coin) to receive online transdiagnostic group CBT in addition to usual postnatal care, or to receive usual postnatal care only.

DETAILED DESCRIPTION:
This study will involve a pilot randomized controlled trial (RCT) to determine the feasibility of a 10-week group CBT intervention for treating postpartum depression and anxiety and study procedures. Primary feasibility objectives include recruitment, completion of study measures, retention and participant satisfaction/acceptability of the intervention. The secondary objective of the pilot RCT is to estimate the treatment effects on PPD and anxiety symptoms to guide the conduct of a future full-scale RCT of the intervention.

48 Participants will be assigned in a 1:1 ratio to the experimental (transdiagnostic CBT group plus treatment as usual (TAU)) or control group (TAU alone). Participants in both groups will complete all study questionnaires at baseline (T1), 10 weeks later (T2 - immediately post-intervention in the experimental group to assess effectiveness), and 6 months after enrollment (T3 - intervention durability). Participants in the treatment group will complete a satisfaction questionnaire with three open-ended questions that will explore their experiences and recommendations for improving the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* have an infant <12 months at recruitment
* fluent in written/spoken English
* have an EPDS score ≥10 and/or a GAD-7 score≥10
* live in Ontario, Canada

Exclusion Criteria:

* does not meet diagnostic criteria for bipolar, psychotic, borderline personality and current substance use disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited in recruitment period | 6 months
  Recruit and randomize 48 participants (over two groups; 24 experimental, 24 control) in six months
Number of participants who complete all data collection procedures | 6 months
  75% of participants complete all three questionnaires and structured interviews
Number of participants who complete study (retention) | 6 months
  75% of participants remain in study until completion
Number of participants who complete the intervention (adherence) | 6 months
  80% of participants in treatment group complete the intervention

SECONDARY OUTCOMES:
Estimate Treatment effect - Edinburgh Postnatal Depression Scale (EPDS) | 10 weeks
  Postpartum depression (PPD) is best conceptualized as a continuous construct with its impact operating across a continuum of severity, and so a continuous measure of PPD (EPDS) is our primary outcome. In keeping with most PPD RCTs, our primary effectiveness timepoint is immediately post-treatment (T2). The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item gold standard measure of PPD. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score of ≥10 is consistent with possible PPD, ≥13 is consistent with probable PPD and changes in scores >4 are accepted as being indicative of clinically significant change.
Estimate Treatment effect - GAD-7 | 10 weeks
  A reliable and valid 7-item self-report scale that assesses the symptoms of generalized anxiety disorder, the most common comorbidity of PPD. A cutoff of ≥10 defines clinically important levels of anxiety symptoms and changes in scores >4 are accepted as being indicative of clinically significant change.

OTHER OUTCOMES:
Parenting Stress Index (PSI-SF) | 10 weeks
  The Parenting Stress Index (short form) is a 36-item parent self-report measure that identifies potentially dysfunctional parent-child systems on three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. The measure also produces a total score that is an indication of overall level of stress a person is feeling in their role as a parent. Higher scores indicate higher levels of stress.
Parenting Stress Index (PSI-SF) | 6 months
  The Parenting Stress Index (short form) is a 36-item parent self-report measure that identifies potentially dysfunctional parent-child systems on three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. The measure also produces a total score that is an indication of overall level of stress a person is feeling in their role as a parent. Higher scores indicate higher levels of stress.
GAD-7 | 6 months
  A reliable and valid 7-item self-report scale that assesses the symptoms of generalized anxiety disorder, the most common comorbidity of PPD. A cutoff of ≥10 defines clinically important levels of anxiety symptoms and changes in scores >4 are accepted as being indicative of clinically significant change.
Multidimensional Scale of Perceived Social Support (MSPSS) | 10 weeks
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
Multidimensional Scale of Perceived Social Support (MSPSS) | 6 months
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
The Postpartum Bonding Questionnaire (PBQ) | 10 weeks
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item maternal-report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
The Postpartum Bonding Questionnaire (PBQ) | 6 months
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item maternal-report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R) | 10 weeks
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R) | 6 months
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
Client Satisfaction Questionnaire (CSQ-8) | 10 weeks
  Intervention participants only. An 8-item scale that measures and assesses consumer satisfaction with health and human services. Items are scored on a 4-point scale and total scores range from 8-32, with higher scores indicating greater satisfaction. Three additional open-ended questions will be asked upon completion of the CSQ-8 to gather feedback from participants in the CBT group about their experience of the intervention and any recommendations they may have for improvement.
Major Depressive Disorder | 10 weeks
  A structured psychiatric interview will assess current psychiatric syndromes in participants. The Diagnostic Assessment Research Tool (DART) will be administered at baseline, 10 weeks, and 6 months to assess change in psychiatric symptoms over the study period.
Major Depressive Disorder | 6 months
  A structured psychiatric interview will assess current psychiatric syndromes in participants. The Diagnostic Assessment Research Tool (DART) will be administered at baseline, 10 weeks, and 6 months to assess change in psychiatric symptoms over the study period.
Edinburgh Postnatal Depression Scale (EPDS) | 6 months
  Postpartum depression (PPD) is best conceptualized as a continuous construct with its impact operating across a continuum of severity, and so a continuous measure of PPD (EPDS) is our primary outcome. In keeping with most PPD RCTs, our primary effectiveness timepoint is immediately post-treatment (T2). The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item gold standard measure of PPD. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score of ≥10 is consistent with possible PPD, ≥13 is consistent with probable PPD and changes in scores >4 are accepted as being indicative of clinically significant change.
Generalized Anxiety Disorder | 10 weeks
  A structured psychiatric interview will assess current psychiatric syndromes in participants. The Diagnostic Assessment Research Tool (DART) will be administered at baseline, 10 weeks, and 6 months to assess change in psychiatric symptoms over the study period.
Generalized Anxiety Disorder | 6 months
  A structured psychiatric interview will assess current psychiatric syndromes in participants. The Diagnostic Assessment Research Tool (DART) will be administered at baseline, 10 weeks, and 6 months to assess change in psychiatric symptoms over the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No